CLINICAL TRIAL: NCT04973267
Title: Game Plan for PrEP: A Pilot Trial of a Web-based Intervention to Help High-risk Men on PrEP Adhere to Their Medication, Reduce Alcohol Use, and Encourage Safe Sex
Brief Title: Game Plan for PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2105002999; 5R34AA027195 (NIH)
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Human Immunodeficiency Virus Exposure; Alcohol; Harmful Use
Keywords: PrEP; Alcohol Use; HIV; STIs; LGBTQ
MeSH Terms: conditions — Alcohol Drinking; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned 1:1 to one of two conditions: (1) Game Plan for PrEP and (2) an attention-matched control consisting of videos encouraging healthy lifestyle habits.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators will be blinded to study condition. Staff collecting dried blood spot samples will also be blinded to condition. Participants will be encouraged to complete online surveys using an automated email system, so outcomes assessors will not be present.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game Plan for PrEP (Experimental): Participants will be asked to use Game Plan for PrEP for however long they wish. Game Plan for PrEP is a web-based intervention that provides users with feedback about how much their risk for HIV is reduced on PrEP, their risk for bacterial STIs, and helps them make a plan to take their medication regularly and reduce their risk for STIs. Game Plan for PrEP also providers users with feedback about their alcohol use compared to others in their age group and encourages them to make a plan to reduce it.
  Interventions: Behavioral: Game Plan for PrEP
- Lifestyle Habits Videos (Sham Comparator): Participants in this condition will view several videos that encourage them to adopt sleep hygiene and healthy diet behaviors. The videos were selected to last as long as the average time users engage with Game Plan for PrEP in its initial modules.
  Interventions: Behavioral: Attention-Matched Control Lifestyle Habits Videos

INTERVENTIONS:
Behavioral: Game Plan for PrEP — See arm description.
  Arms: Game Plan for PrEP
Behavioral: Attention-Matched Control Lifestyle Habits Videos — Web-based videos providing information on sleep hygiene and proper diet.
  Arms: Lifestyle Habits Videos

SUMMARY:
This small pilot randomized controlled trial will test whether a brief, web-based intervention inspired by the principles of motivational interviewing helps high-risk men who take pre-exposure prophylaxis (PrEP) moderate their alcohol use, and improve key outcomes of PrEP care, including adherence, persistence, and STI rates. Men with a history of "lapses" in PrEP adherence will be randomly assigned to either (1) use the web-based intervention, called Game Plan for PrEP, or (2) watch video clips encouraging healthy lifestyles (e.g., sleep hygiene, balanced diet; attention-matched control). Participants will complete STI testing and submit dried blood spot (DBS) samples to facilitate analyses of alcohol use and PrEP adherence biomarkers at baseline, 3-months, and 6-months during the study period. Participants will also complete online surveys at baseline, 1-month, 3-months, and 6-months during the study period.

DETAILED DESCRIPTION:
This small, pilot randomized controlled trial will explore preliminary evidence for the efficacy of Game Plan for PrEP, a brief, web-based intervention inspired by brief motivational interventions. The study will test whether Game Plan for PrEP is efficacious in reducing heavy drinking and sexually-transmitted infection (STI) incidence, and improving PrEP adherence/persistence, among heavy drinking men who have sex with men who are on PrEP, but who report a recent history of missing 3 or more consecutive doses in the past month. In this study, we will randomize 50 gay and bisexual men to receive either (1) Game Plan for PrEP (GP4PrEP) or (2) an attention-matched control at the same PrEP care/monitoring visit that they reported meeting eligibility criteria. We will use self-report measures of alcohol use collected at 1-, 3-, and 6-months and changes in a biomarker of alcohol use collected at baseline, 3-, and 6-months to explore whether Game Plan for PrEP reduces binge drinking compared with control. We will also use data from a biomarker of PrEP adherence to explore whether Game Plan for PrEP improves PrEP adherence versus control.

ELIGIBILITY:
Inclusion Criteria:

* Current male gender
* 18+ years old
* Fluent in English
* Heavy alcohol use in the past month (>5 drinks on a single occasion or >14 drinks in a week)
* Currently prescribed and actively taking PrEP
* Report missing > 3 PrEP doses in a row at least once in the past 3 months.

Exclusion Criteria:

* Reporting a history or risk of complicated alcohol withdrawal
* Reporting currently receiving medications or counseling for an alcohol or drug use disorder
* Injection drug use in the past year
* Positive screen for drug-related disorders

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants will be assigned male sex at birth and report current male gender.
Enrollment: 73 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Wray, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants will be asked to use Game Plan for PrEP for however long they wish. Game Plan for PrEP is a web-based intervention that provides users with feedback about how much their risk for HIV is reduced on PrEP, their risk for bacterial STIs, and helps them make a plan to take their medication regularly and reduce their risk for STIs. Game Plan for PrEP also providers users with feedback about their alcohol use compared to others in their age group and encourages them to make a plan to reduce it.
- Control: Participants in this condition will view several videos that encourage them to adopt sleep hygiene and healthy diet behaviors. The videos were selected to last as long as the average time users engage with Game Plan for PrEP in its initial modules.
  Attention-Matched Control Lifestyle Habits Videos: Web-based videos providing information on sleep hygiene and proper diet.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 37 | 36
Completed | 37 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (7.4) | 37.4 (10) | 35.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 37 | 36 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 30 | 30 | 60
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Years on PrEP [Mean (Standard Deviation); unit: years] | 2.7 (2.2) | 2.5 (2.2) | 2.6 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Pre-exposure Prophylaxis (PrEP) Lapse Days
Description: Number of participants who reported missing 4+ consecutive days of PrEP doses
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 36
Participants | 3 | 3

2. Primary Outcome: Persistence With Pre-exposure Prophylaxis (PrEP)
Description: Whether or not participants explicitly stopped taking PrEP at some point during the 6-month study period
Time Frame: Past 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 36
Participants | 5 | 7

3. Primary Outcome: Number of Alcohol Drinking Days
Description: The total number of days in which participants reported drinking alcohol in the past 30 days
Time Frame: Month 1, Month 3, and Month 6
Measure: Mean (Standard Error); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 36
days
  Month 1 | 9.98 (1.29) | 11.38 (1.49)
  Month 3 | 9.12 (1.20) | 7.49 (1.03)
  Month 6 | 7.21 (0.97) | 9.25 (1.28)

4. Primary Outcome: Average Number of Drinks Consumed Per Drinking Day
Description: The average number of standard alcoholic drinks consumed when participants reported drinking over the past 30 days
Time Frame: Month 1, Month 3, and Month 6
Measure: Mean (Standard Error); unit: standard drinks
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 36
standard drinks
  Month 1 | 3.89 (0.36) | 4.02 (0.37)
  Month 3 | 4.37 (0.37) | 4.60 (0.37)
  Month 6 | 3.94 (0.37) | 4.49 (0.40)

5. Primary Outcome: Number of Heavy Drinking Days (5+ Drinks on a Single Occasion)
Description: The total number of days on which participants reported drinking 5+ drinks in a single day over the past 30 days
Time Frame: Month 1, Month 3, and Month 6
Measure: Mean (Standard Error); unit: bring drinking days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 36
bring drinking days
  Month 1 | 2.70 (0.54) | 3.84 (0.70)
  Month 3 | 2.70 (0.55) | 2.58 (0.50)
  Month 6 | 2.82 (0.57) | 3.65 (0.71)

6. Secondary Outcome: Phosphatidylethanol Level
Description: The quantity of phosphatidylethanol (PEth) detected in dried blood spot samples collected at 3- and 6-months, ng/mL
Time Frame: Month 3 and Month 6
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 36
ng/mL
  Month 3 | 95.57 (8.03) | 77.61 (8.59)
  Month 6 | 72.47 (8.79) | 93.58 (9.49)

7. Secondary Outcome: Tenofovir Diphosphate Adherence
Description: The predicted probability of tenofovir diphosphate adherence (>= 4 doses/week) detected in dried blood spot samples collected at 3- and 6-months
Time Frame: Month 3 and Month 6
Measure: Mean (Standard Error); unit: predicted probability
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 36
predicted probability
  Month 3 | 0.68 (0.09) | 0.83 (0.07)
  Month 6 | 0.76 (0.08) | 0.74 (0.08)

8. Secondary Outcome: Any Sexually-transmitted Infection (STI) Diagnosis
Time Frame: 6 Months
Population: No data were collected
Arm/Group | Game Plan for PrEP | Lifestyle Habits Videos
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 0/37 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT04973267/Prot_000.pdf
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT04973267/ICF_001.pdf